CLINICAL TRIAL: NCT03325738
Title: Cetuximab for Unresectable Cutaneous Squamous Cell Carcinoma - A National Retrospective Study
Acronym: C3
Status: Completed | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/05
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Squamous Cell Cutaneous Carcinoma of the Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Localized cutaneous squamous cell carcinoma (CSCC) is usually treated by radical surgery with or without radiotherapy. The cure rate is high around 90% of cases (1). Unresectable CSCC represents less than 10% of all CSCC. The prognosis of these advanced forms is poor, without any proven treatment option. The number of studies investigating systemic treatment of advanced or metastatic CSCC is limited, mostly based on phase II trials or case reports. Systemic treatment includes cytotoxic chemotherapy such as cisplatin and 5-Fluoro-uracil (5FU), immunotherapy (interferon alpha) or retinoic acid (13CRa) (1,2). Recently, epidermal growth factor receptor (EGFR) targeting agents have been explored (1,2). The anti-EGFR monoclonal antibody Cetuximab has shown some clinical efficacy in advanced CSCC alone or concomitant with radiotherapy or chemotherapy (3-5). A recent phase II study aimed at investigating the role of Cetuximab in 36 patients with unresectable CSCC (6). The authors reported a disease control rate at 6 weeks of 69% (95% CI, 52% to 84%). The best responses were eight partial responses and two complete responses. There were no Cetuximab-related deaths. There were three related serious adverse events: two grade 4 infusion reactions and one grade 3 interstitial pneumopathy. Grade 1 to 2 acne-like rash occurred in 78% of patients and was associated with prolonged Progression Free Survival (PFS) (6). The authors concluded that regarding the Cetuximab therapeutic index it could be interesting in this particular situation mainly for elderly patient. Unfortunately, the small number of patient included not allowed to draw definitive conclusion. It was interesting to note that the Disease rate control (DRC) with Cetuximab increased of 15% comparatively of DRC with chemotherapy. Additionally it seems that in case of efficacy the functional improvement of Cetuximab-sensitive patients occurred after very few infusions.

Taking these data together it seemed logical to design a larger retrospective clinical trial to confirm these results in "real life patients".

ELIGIBILITY:
Inclusion Criteria

1. Histologically Confirmed squamous cell cutaneous carcinoma of the skin (SCCS)
2. Locally advanced SCCS that is surgically unresectable, or metastatic SCCS, with documented progression, and who received a treatment of Cetuximab in monotherapy,
3. Patients have to be anti EGFR-naïve,
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group performance status ≤ 2; life expectancy ≥ 3 months
6. Presence of at least one measurable target lesion, according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
7. Adequate hematologic, hepatic, and renal functions
8. Available medical data
9. Chemotherapy naïve patient in metastatic or locally advanced conditions (Cisplatinum used concomitantly with radiotherapy is allowed)

Exclusion criteria

1. Prior radiotherapy within the last 4 weeks before the start of cetuximab (radiotherapy in concomitance with cetuximab is allowed if this is administrated in another lesion than the lesion treated by Cetuximab).
2. Prior therapy with an agent that targets EGFR
3. Instable systemic diseases or active uncontrolled infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a confirmed squamous cell cutaneous carcinoma of the skin, locally Advanced or metastatic and who received a monotherapy treatment by cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit of Cetuximab at 6 weeks | 6 weeks
  To Assess the clinical benefit (complete response [CR], partial response [PR], or stable disease [SD]) after 6 weeks of treatment with Cetuximab

SECONDARY OUTCOMES:
Objective response rate ORR | December 2017
  The ORR will be defined as the sum of partial responses plus complete responses after 6 weeks of treatment with Cetuximab.
Overall survival OS | December 2017
  2. The OS will be calculated between date of treatment beginning (Cetuximab) and the date of death for any reason. Patients who did not die at the time of analysis or are lost of follow-up will be censored at the date of the latest news.
Progression free survival PFS | December 2017
  The PFS will be calculated between date of treatment beginning (Cetuximab) and date of progression, death or starting another anticancer treatment. Patients who did not progress, did not die at the time of analysis or are lost of follow-up will be censored at the date of the latest news.
Cetuximab safety | December 2017
  The safety profile will be described using the common toxicity criteria from the NCI v4.03 and biological, including occurrence of acne-like rash.
Overall response delay | December 2017
  The DOR will be measured from the time measurement criteria are first met for CR/PR until the first date that progressive disease is objectively documented (without other anticancer treatment).
Disease stabilization delay | December 2017
  The DSD will be measured from the start of the treatment until the criteria for progression is objectively documented.
Best overall response BOR | December 2017
  The BOR will be recorded from the start of the treatment until the end of treatment taking into account any requirement for confirmation.

CONTACTS AND LOCATIONS:
Locations (1):
- PEYRADE Frédéric, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided